CLINICAL TRIAL: NCT02334969
Title: A Multi-center, Randomized, Double-blind and Placebo-controlled Clinical Research of 2200 Cases in Improving Curative Effect of Secondary Prevention for Patients With Ischemic Stroke Through Syndrome Differentiation of TCM
Brief Title: Curative Efficacy of Secondary Prevention for Patients With Ischemic Stroke Through Syndrome Differentiation of TCM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xiaofei Yu (Other)
Collaborators: Shanghai Municipal Science and Technology Commission (Other Government)
Responsible Party: Sponsor-Investigator, Xiaofei Yu, Shuguang Hospital, ShuGuang Hospital
Organization: ShuGuang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 14401970300
Record Dates: First submitted 2015-01-06; First posted 2015-01-09 (Estimated); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Ischemic Stroke
Keywords: ischemic stroke；Naoxintong Capsule
MeSH Terms: conditions — Ischemic Stroke | interventions — naoxintong

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental group (Experimental): On the basis of the secondary prevention of ischemic stroke，Volunteers will be taken Naoxintong capsule, 2 times a day, three granule per time
  Interventions: Drug: Naoxintong Capsule
- Control group (Active Comparator): On the basis of the secondary prevention of ischemic stroke，Volunteers will be taken Placebo capsule，which is identical with Naoxintong capsule in the appearance, shape, color and content, 2 times a day, three granule per time
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naoxintong Capsule — This is Naoxintong capsule,which is composed of Huangqi,Chishao,Danshen,Danggui, Chuanxiong,Taoren,Honghua,Ruxiang,Moyao,Jixueteng,Niuxi,Guizhi,Sangzhi,Dilong,Quanxie,etal.
  Other Names: Chinese Herbal Compound
  Arms: Experimental group
Drug: Placebo — placebo capsule has the same as Naoxintong capsule in the appearance, shape,colour and content tinct.
  Other Names: Placebo of Chinese Herbal Compound
  Arms: Control group

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Naoxintong Capsule in the secondary prevention of ischemic stroke by the multi-center, randomized,double-blind，placebo-controlled trial design project.

DETAILED DESCRIPTION:
The research employs a random, double-blind, multicenter, placebo parallel and controlled design to observe the clinical effect of Naoxintong capsule in the treatment in ischemic stroke of the blood stasis syndrome on the secondary prevention，which is funded by Science and Technology Commission of Shanghai Municipality.The therapeutic drug of the research is Naoxintong capsule on the market for treatment and prevention of stroke, applicable to stroke patients caused by qi deficiency, blood stasis and venation stasis.The research will be carried out in 24 hospitals.It is a total number of 2200 volunteers，who will meet the inclusion criteria other than the exclusion criteria and agree to participate in the research.Volunteers will be randomly assigned to the experimental group or the control group. The trial drug for the experimental group is Naoxintong capsule, while that for the control group is a kind of placebo capsule.Volunteers will be regularly followed up during the experimental period of 2 years. It will be to evaluate the clinical efficacy of Naoxintong capsule on the secondary prevention by the stroke recurrence and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Adult volunteers aged ≤ 90 years old, ≥18 years old；
* Conforming to the diagnostic criteria of cerebral infarction under the 2010 version of Chinese Guidelines for Treatment of Acute Ischemic Stroke；
* Conforming to diagnostic criteria of the stasis type of TCM on the ischemic stroke；
* The onset of acute cerebral infarction ≥ 10 days；
* Consciousness awake；
* Volunteers agree to accept the program and sign informed consent.

Exclusion Criteria:

* Excluding the patients of the yin deficiency type of ischemic stroke.The diagnostic criteria of Yin deficiency type of ischemic stroke is that sudden onset of disease；being signs or symptoms of of neurological deficit；CT or MRI examination showing intracranial ischemic lesions；Scarlet tongue；
* The volunteers with severe heart diseases, cardiac insufficiency, hepatosis, renal insufficiency, respiratory failure, malignant tumour, alimentary tract hemorrhage, etc. who may fail to complete the two-year follow-up；
* Psychiatric patients；
* Pregnants and lactating women；
* Volunteers in other clinical trials；
* Volunteers who are not suitable for this clinical trial according to the researchers for other reasons.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2200 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Stroke recurrence rate and Stroke mortality | 2 years
  Stroke recurrence rate and Stroke mortality

SECONDARY OUTCOMES:
All-cause mortality | 2 years
  All-cause mortality
The incidence rate of myocardial infarction | 2 years
  The incidence rate of myocardial infarction

OTHER OUTCOMES:
The incidence of adverse events | 2 years
  The incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Xiao F Yu, Doctor, Study Chair — ShuGuang Hospital
Locations (24):
- China (24):
  - Shanghai seventh People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Ninth People's Hospital affliated to Shanghai Jiao Tong University Shool of Medcine, Shanghai, Shanghai Municipality
  - North Branch of Ruijin Hospital affliated to Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Shanghai Putuo Central Hospital, Shanghai, Shanghai Municipality
  - Shuguang Hospital affliated to Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Longhua Hospital affliated to Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Zhongshan Hospital affliated to Fudan University, Shanghai, Shanghai Municipality
  - Huashan Hospital affliated to Fudan University, Shanghai, Shanghai Municipality
  - Shanghai fifth People's Hospital affliated to Fudan University, Shanghai, Shanghai Municipality
  - Tongren Hospital affliated to Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Tongji Hospital, Shanghai, Shanghai Municipality
  - Shanghai Chinese Medicine Hospital, Shanghai, Shanghai Municipality
  - Shanghai tenth People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Hospital of Integrative Medicine, Shanghai, Shanghai Municipality
  - Xinhua Hospital affliated to Shanghai Jiao Tong University Shool of Medcine, Shanghai, Shanghai Municipality
  - Dongfang Hospital affliated to Tongji University, Shanghai, Shanghai Municipality
  - Pudong Gong Li Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Shanghai sixth People's Hospital affliated to Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Changning Tongren Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Changhai Hospital, Shanghai, Shanghai Municipality
  - Pudong Hospital of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - East Branch of Shanghai sixth People's Hospital, Shanghai, Shanghai Municipality
  - Qingpu Branch of Zhongshan Hospital affliated to Fudan University, Shanghai, Shanghai Municipality
  - Shanghai third People's Hospital affliated to Shanghai Jiao Tong University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Antithrombotic Trialists' Collaboration. Collaborative meta-analysis of randomised trials of antiplatelet therapy for prevention of death, myocardial infarction, and stroke in high risk patients. BMJ. 2002 Jan 12;324(7329):71-86. doi: 10.1136/bmj.324.7329.71. PMID 11786451
- [Result] Hankey GJ. Ischaemic stroke--prevention is better than cure. J R Coll Physicians Edinb. 2010 Mar;40(1):56-63. doi: 10.4997/JRCPE.2010.111. No abstract available. PMID 21125042
- [Result] Sobel M. Commentary. Aspirin plus dipyridamole versus aspirin alone after cerebral ischaemia of arterial origin (ESPRIT): randomised controlled trial. Perspect Vasc Surg Endovasc Ther. 2007 Mar;19(1):87-9. doi: 10.1177/1531003507299489. No abstract available. PMID 17437989
- [Result] Matchar DB, Samsa GP, Liu S. Cost-effectiveness of antiplatelet agents in secondary stroke prevention: the limits of certainty. Value Health. 2005 Sep-Oct;8(5):572-80. doi: 10.1111/j.1524-4733.2005.00050.x. PMID 16176495
- [Result] Diener HC, Sacco RL, Yusuf S, Cotton D, Ounpuu S, Lawton WA, Palesch Y, Martin RH, Albers GW, Bath P, Bornstein N, Chan BP, Chen ST, Cunha L, Dahlof B, De Keyser J, Donnan GA, Estol C, Gorelick P, Gu V, Hermansson K, Hilbrich L, Kaste M, Lu C, Machnig T, Pais P, Roberts R, Skvortsova V, Teal P, Toni D, VanderMaelen C, Voigt T, Weber M, Yoon BW; Prevention Regimen for Effectively Avoiding Second Strokes (PRoFESS) study group. Effects of aspirin plus extended-release dipyridamole versus clopidogrel and telmisartan on disability and cognitive function after recurrent stroke in patients with ischaemic stroke in the Prevention Regimen for Effectively Avoiding Second Strokes (PRoFESS) trial: a double-blind, active and placebo-controlled study. Lancet Neurol. 2008 Oct;7(10):875-84. doi: 10.1016/S1474-4422(08)70198-4. Epub 2008 Aug 29. PMID 18757238
- [Result] Uchiyama S, Ikeda Y, Urano Y, Horie Y, Yamaguchi T. The Japanese aggrenox (extended-release dipyridamole plus aspirin) stroke prevention versus aspirin programme (JASAP) study: a randomized, double-blind, controlled trial. Cerebrovasc Dis. 2011;31(6):601-13. doi: 10.1159/000327035. Epub 2011 Apr 19. PMID 21502757
- [Result] Jeng JS, Sun Y, Lee JT, Lin RT, Chen CH, Po HL, Lin HJ, Liu CH, Sun MH, Sun MC, Chern CM, Lien LM, Chiu HC, Hu HH, Chiou HY, Chen ST, Ma H, Hsu CY; SPAD Study Investigators. The efficacy and safety of cilostazol in ischemic stroke patients with peripheral arterial disease (SPAD): protocol of a randomized, double-blind, placebo-controlled multicenter trial. Int J Stroke. 2015 Jan;10(1):123-7. doi: 10.1111/ijs.12384. Epub 2014 Nov 14. PMID 25394855
- [Result] Ikeda Y, Shimada K, Teramoto T, Uchiyama S, Yamazaki T, Oikawa S, Sugawara M, Ando K, Murata M, Yokoyama K, Ishizuka N. Low-dose aspirin for primary prevention of cardiovascular events in Japanese patients 60 years or older with atherosclerotic risk factors: a randomized clinical trial. JAMA. 2014 Dec 17;312(23):2510-20. doi: 10.1001/jama.2014.15690. PMID 25401325
- [Derived] Yu XF, Zhu XY, Yuan CX, Wu DH, Zhao YW, Yang JJ, Wang CD, Wu WW, Liu XY, Liu ZG, Nie ZY, Deng BQ, Bao H, Li LX, Wang CY, Zhang HZ, Zhang JS, Huang JH, Gong F, Wang MZ, Guo YM, Sun Y, Cai DF. Naoxintong Capsule for Secondary Prevention of Ischemic Stroke: A Multicenter, Randomized, and Placebo-Controlled Trial. Chin J Integr Med. 2022 Dec;28(12):1063-1071. doi: 10.1007/s11655-022-3586-8. Epub 2022 Oct 17. PMID 36251140